CLINICAL TRIAL: NCT01230580
Title: A Randomised Controlled Trial of a Strategy of Switching to Boosted PI Monotherapy Versus Continuing Combination ART for the Long-term Management of HIV-1 Infected Patients Who Have Achieved Sustained Virological Suppression on HAART
Brief Title: Protease Inhibitor Monotherapy Versus Ongoing Triple-therapy in the Long Term Management of HIV Infection (PIVOT)
Acronym: PIVOT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical Research Council (Other Government)
Collaborators: NHS Health Technology Assessment Programme (Other)
Responsible Party: Medical Research Council (Dr Nick Paton Chief Investigator MRC Clinical Trials Unit), Medical Research Council
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PIVOT; 2007-006448-23 (EudraCT Number)
Record Dates: First submitted 2010-10-27; First posted 2010-10-29 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2010-10

CONDITIONS: HIV Infection; Acquired Immunodeficiency Syndrome
Keywords: Protease Inhibitors; RNA virus infections; Virus diseases; Sexually Transmitted Diseases viral; Immune system diseases; Anti-infective Agents; Drug resistance
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; RNA Virus Infections; Virus Diseases; Sexually Transmitted Diseases, Viral; Immune System Diseases | interventions — Protease Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Protease Inhibitor Monotherapy (Experimental): Ritonavir-boosted protease inhibitor
  Interventions: Drug: Protease Inhibitor
- Control (Active Comparator): Standard-of-care triple-therapy regimen
  Interventions: Drug: Standard-of-care Antiretroviral therapy

INTERVENTIONS:
Drug: Protease Inhibitor — Switch to a regimen comprising a single ritonavir-boosted Protease Inhibitor
  Arms: Protease Inhibitor Monotherapy
Drug: Standard-of-care Antiretroviral therapy — Regimen should consist of 3 drugs: 2 nucleoside reverse transcriptase inhibitors with either a non-nucleoside reverse transcriptase inhibitor or a protease inhibitor
  Arms: Control

SUMMARY:
The PIVOT trial aims to determine whether a strategy of switching to PI monotherapy is non-inferior to continuing triple-therapy, in terms of the proportion of patients who maintain all the drug treatment options that were available to them at baseline after at least 3 years of follow-up, and to compare clinical events, safety, toxicity and health economic parameters between the two strategies.

ELIGIBILITY:
Inclusion Criteria:

Vl < 50 for 24 weeks prior to screening CD4 > 100 at screening

Exclusion Criteria:

1. Known major protease resistance mutation(s) documented on prior resistance testing if performed (prior resistance testing is not mandatory for trial participation).
2. Previous change in ART drug regimen for reasons of unsatisfactory virological response (patients who have changed regimen for prevention or management of toxicity or to improve regimen convenience are permitted to enter the trial).
3. Previous allergic reaction to a PI.
4. Patient currently using or likely to require use of concomitant medication with known interaction with PIs.
5. Patient requiring treatment with radiotherapy, cytotoxic chemotherapy, or is anticipated to need these during the trial period.
6. Treatment for acute opportunistic infection within 3 months prior to trial screening.
7. Pregnant or trying to become pregnant at the time of trial entry.
8. History of active substance abuse or psychiatric illness that, in the opinion of the investigator, would preclude compliance with the protocol, dosing schedule or assessments.
9. History of HIV encephalopathy with current deficit >1 in any domain of the Neuropsychiatric AIDS Rating Scale (see Appendix 7).
10. Past or current history of cardiovascular disease, or 10 year absolute coronary heart disease risk of >30%, or risk of >20% if the patient has diabetes or a family history of premature ischaemic heart disease or stroke.
11. History of insulin-dependent diabetes mellitus.
12. Patient currently receiving interferon therapy for Hepatitis C virus infection or planning to start treatment for Hepatitis C at the time of trial entry.
13. Co-infection with hepatitis B, defined as Hepatitis BsAg positive at screening or at any time since HIV diagnosis, unless the patient has had a documented Hepatitis B DNA measurement of less than 1000 copies/ml taken whilst off Hepatitis B active drugs.
14. Any other active clinically significant condition, or findings during screening medical history or examination, or abnormality on screening laboratory blood tests that would, in the opinion of the investigator, compromise the patient's safety or outcome in the trial.
15. Fasting plasma glucose >7.0mmol/L at trial screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 587 (Actual)
Dates: Start 2008-11; Primary Completion 2013-11 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Loss of future drug options | Up to 5 years
  The first occurrence of intermediate to high level resistance to any one or more of the standard antiretroviral drugs (limited to licensed drugs in contemporary use) to which the patient's virus was considered to be sensitive at trial entry (i.e. excluding drug resistance that was known to be present on previous resistance testing).

SECONDARY OUTCOMES:
Death from any cause | Up to 5 years
Serious AIDS-defining illness | Up to 5 years
Serious non-AIDS defining illness | Up to 5 years
Adverse events | Up to 5 years
Confirmed Virological rebound | Up to 5 years
CD4+ count change | Up to 5 years
Health-related Quality of Life change | Up to 5 years
Neurocognitive function change | Up to 5 years
Cardiovascular risk change | Up to 5 years
Health care costs | Up to 5 years
HIV VL in Genital Secretions | Week 96
  In a sub-set of participants (n=73):-
  * Compare prevalence of detectable VL and magnitude of viral replication in genital secretions in patients taking PI monotherapy and triple therapy; to test if PI monotherapy is non-inferior to triple therapy.
  * Compare drug levels in genital secretions and plasma.
  * Describe the profile of drug resistance (if any) in patients with detectable VL in genital secretions and to compare this with any previous or subsequent resistance profile in plasma.
  (Genital Secretions substudy REC # 09/H0305/58)
HIV VL in CSF | Week 96
  In a subset of participants on PI monotherapy (n=40).
  * Estimate the proportion of patients who have detectable HIV viral load in CSF after 48 weeks on PI monotherapy, and to refute the hypothesis that this proportion is greater than 20%.
  * Assess whether CSF markers of CNS immune activation, inflammation and neuronal degeneration are elevated after 48 weeks on PI monotherapy.
  * Assess whether CSF HIV viral load and markers of immune activation, inflammation and neuronal degeneration are elevated in patients with symptomatic CNS disease.
  (CNS substudy REC # 09/H0305/58).

CONTACTS AND LOCATIONS:
Overall Officials: Nick Paton, MD, Principal Investigator — Medical Research Council

REFERENCES:
- [Derived] Winston A, Arenas-Pinto A, Stohr W, Fisher M, Orkin CM, Aderogba K, De Burgh-Thomas A, O'Farrell N, Lacey CJ, Leen C, Dunn D, Paton NI; PIVOT Trial Team. Neurocognitive function in HIV infected patients on antiretroviral therapy. PLoS One. 2013 Apr 30;8(4):e61949. doi: 10.1371/journal.pone.0061949. Print 2013. PMID 23646111